CLINICAL TRIAL: NCT01017562
Title: Differentiation of Aseptic From Septic Loosening in Patients With Total Hip Arthroplasty Using 18F-fluoride PET
Brief Title: Differentiation of Aseptic From Septic Loosening by 18F-fluoride PET
Status: Completed | Type: Observational
Sponsor: Yokohama City University Medical Center (Other)
Other Study IDs: YCU21-106
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Hip Arthroplasty
Keywords: To clarify the 18F-fluoride uptake patterns associated with aseptic or septic loosening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- condition of joint implant

SUMMARY:
In this study, the investigators utilized the 18F-fluoride PET method to evaluate THA cases with a stable, septic or septic loosened implant in order to differentiate these clinical settings using a novel uptake type classification approach.

ELIGIBILITY:
Exclusion Criteria:

* Within one year after surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients after total hip arthroplasty who agreed with the informed consent for this study.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2007-04; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Kobayashi, MD, PhD., Principal Investigator — Department of orthopaedic surgey, Yokohama City University
Locations (1):
- Departement of orthopaedic sugery, Yokohama, Kanagawa, Japan